CLINICAL TRIAL: NCT06367530
Title: Global Survey of Trilateral Retinoblastoma: Incidence and Outcomes
Brief Title: Trilateral Retinoblastoma: Incidence and Outcomes
Acronym: GS-TRIO
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Marcus de Jong, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: GS-TRIO-2024
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Trilateral Retinoblastoma; Retinoblastoma
Keywords: survival; trilateral retinoblastoma; retinoblastoma; incidence; global
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Incidence and survival of trilateral retinoblastoma and the differences globally — The detection and survival of trilateral retinoblastoma around the world and for instance differences between high- and low-income countries in terms of incidence and survival.

SUMMARY:
Patients with heritable retinoblastoma are at risk to develop an intracranial brain tumor, which is often fatal. The investigators intend to look at the incidence and survival of trilateral retinoblastoma (which is a brain tumor that can either be located in the pineal gland or elsewhere in the brain) in retinoblastoma patients globally. All retinoblastoma patients from participating centers will be included. The investigators hypothesize that the apparent incidence of trilateral retinoblastoma (especially the usually later diagnosed pineal trilateral retinoblastoma) in low-income countries will be lower because of low chances of surviving the ocular tumors at about 50% and also because of possible under-diagnosis. Therefore, as retinoblastoma care improves in low-income countries the incidence of (pineal) trilateral retinoblastoma might go up. Knowledge about incidence and survival can help improve health practices in parts of the world where this might be needed. Therefore this global study firstly aims 1) to evaluate survival after trilateral retinoblastoma and factors influencing survival and 2) to evaluate incidence of trilateral retinoblastoma by country income level. The study will run from 2024 through 2027.

DETAILED DESCRIPTION:
This study will adhere to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement for cohort studies and to the Guidelines for Accurate and Transparent Health Estimates Reporting (GATHER) statement. The study is designed as a prospective cohort study of retinoblastoma patients diagnosed in one year from as many as possible worldwide treatment centers. The methods of patient recruitment are partly similar to previous global retinoblastoma studies. Data will be extracted from a the Global Retinoblastoma study follows up patients who will present with retinoblastoma in 2024-2027.

All unique trilateral retinoblastoma patients (cases) and all other retinoblastoma patients (controls) with will be included in the incidence analysis. For survival analysis follow-up data will be required.

After initial submission of case data by participating centers three years after the start of the study information on follow-up, metastasis, eye globe salvage, laterality, diagnosis of trilateral retinoblastoma and survival outcome will be available. At a later stage participating centers that reported trilateral retinoblastoma cases will be contacted again for additional information. All trilateral retinoblastoma patients will be included in the analysis, regardless if additional information is provided.

The investigators will request the following additional data:

* location (pineal, supra-/parasellar, other location (e.g., 3rd ventricle)),
* treatment for trilateral retinoblastoma,
* if not clear from initial report: cause of death (trilateral retinoblastoma, side effect of treatment, other),
* details on (germline) RB1 mutation.
* country of residence,
* family history of retinoblastoma,
* was patient symptomatic or asymptomatic when trilateral retinoblastoma was diagnosed (if symptomatic: what where the symptoms? If asymptomatic: how was the tumor diagnosed),
* information on trilateral retinoblastoma confirmation (e.g., biopsy, CSF, treatment response, disease progression),
* treatment for trilateral retinoblastoma,
* was the treatment with intent to cure (active treatment) or was the intent palliative,
* maximum diameter (mm) of tumor,
* wat trilateral retinoblastoma metastasized at the time of diagnosis,
* was this case published (if yes: where?),
* also missing data during the initial submission phase will be requested again.

If feasible additionally all centers that will also be asked if they can retrospectively provide data on trilateral retinoblastoma patients of whom retinoblastoma was not diagnosed in 2024 and were diagnosed with trilateral retinoblastoma in the years 2020 through 2027.

Outcome measures

Incidence and risk factors of developing trilateral retinoblastoma will be analyzed in the following manner (cases and controls who were diagnosed with retinoblastoma in 2024):

* overall incidence of pineal and non-pineal trilateral retinoblastoma in all retinoblastoma patients, bilateral retinoblastoma patients and heritable retinoblastoma patients (all patients with wither bi- or trilateral retinoblastoma, familial retinoblastoma or a proven germline RB1 mutation will be considered heritable),
* estimate possible under-diagnosis of trilateral retinoblastoma in lower-income countries,
* potential modifiers of incidence (risk of developing trilateral retinoblastoma) will be analyzed: pineal versus non-pineal trilateral retinoblastoma, age at diagnosis of retinoblastoma (e.g., < or ≥ 12 months old), country income level.

Survival analysis of trilateral retinoblastoma alone (all cases who were diagnosed with trilateral retinoblastoma in the years 2024 through 2027):

* overall and trilateral retinoblastoma specific survival will be analyzed,
* potential predictors of survival (e.g., pineal versus non-pineal trilateral retinoblastoma, tumor size, previous treatment for retinoblastoma, treatment for trilateral retinoblastoma, symptomatic versus asymptomatic, RB1 mutation, active treatment, metastastic disease, country income level).

Survival analysis of trilateral retinoblastoma in the entire retinoblastoma cohort (cases and controls who were diagnosed with retinoblastoma in 2024-2027):

* trilateral retinoblastoma mortality versus other-cause mortality (also stratified by country income level and al versus non-pineal trilateral retinoblastoma),
* event-free survival (with an event defined as trilateral retinoblastoma diagnosis) (also stratified by country income level and al versus non-pineal trilateral retinoblastoma),
* event-free survival will be analyzed for potential predictors (age at diagnosis of retinoblastoma, previous systemic chemotherapy, previous external beam radiotherapy, country income level).

Other analyses (all cases who were diagnosed with trilateral retinoblastoma in the years 2024 through 2027):

* verify independence between the age at diagnosis of retinoblastoma and trilateral retinoblastoma,
* verify the period that retinoblastoma patients are at risk to develop trilateral retinoblastoma,
* whether trilateral retinoblastoma is usually diagnosed at a later date if the diagnosis of retinoblastoma was before the age of 12 months,
* evaluate and more precisely estimate of the previously estimated lead time between symptomatic and asymptomatic trilateral retinoblastoma of about 1 year.

The income level of a country will be determined by the at the time most recent World Population Prospects by the Department of Economic and Social Affairs of the United Nations.

Statistical analysis

Incidence will be reported as proportions with 95% exact binomial confidence intervals. Cumulative incidence of trilateral retinoblastoma curves will be created, accounting for death from other causes without diagnosis of trilateral retinoblastoma.

Overall survival (all-cause mortality), disease specific survival and event free survival were performed. An event is defined as being diagnosed with trilateral retinoblastoma.

The Kaplan-Meier product-limit method and the log rank test will be used to analyze survival data. A Cox proportional hazards model will be employed to analyze potential predictors factors. Schoenfeld residuals will be used to check the proportionality assumption of the model.

The investigators each case with a unique identifier for stratification based on the center to account for heterogeneity between these centers.

In case of subgroup analyses original P-values will presented, as well as adjusted p-values corrected for multiple hypothesis testing according to Bonferroni's method.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with retinoblastoma

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As many centers in the world will be/have been contacted to participate in this study to provide information about their population of retinoblastoma and trilateral retinoblastoma patients. This study will come as close as possible to an overview of this disease worldwide.
Sampling Method: Probability Sample
Enrollment: 4351 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants (retinoblastoma patients) that will be diagnosed with trilateral retinoblastoma (incidence) | 6 years
  The proportion of patients that be diagnosed with trilateral retinoblastoma in the included cohort of retinoblastoma patients
Overall and event-free survival after being diagnosed with trilateral retinoblastoma | 6 years
  The overall and event free survival of patients diagnosed with trilateral retinoblastoma in the included cohort of retinoblastoma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus de Jong, MD PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
This decision depends on the policy of the the global retinoblastoma study 2024-2027.

REFERENCES:
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Result] Stevens GA, Alkema L, Black RE, Boerma JT, Collins GS, Ezzati M, Grove JT, Hogan DR, Hogan MC, Horton R, Lawn JE, Marusic A, Mathers CD, Murray CJ, Rudan I, Salomon JA, Simpson PJ, Vos T, Welch V; (The GATHER Working Group). Guidelines for Accurate and Transparent Health Estimates Reporting: the GATHER statement. Lancet. 2016 Dec 10;388(10062):e19-e23. doi: 10.1016/S0140-6736(16)30388-9. Epub 2016 Jun 28. PMID 27371184
- [Result] Global Retinoblastoma Study Group; Fabian ID, Abdallah E, Abdullahi SU, Abdulqader RA, Adamou Boubacar S, Ademola-Popoola DS, Adio A, Afshar AR, Aggarwal P, Aghaji AE, Ahmad A, Akib MNR, Al Harby L, Al Ani MH, Alakbarova A, Portabella SA, Al-Badri SAF, Alcasabas APA, Al-Dahmash SA, Alejos A, Alemany-Rubio E, Alfa Bio AI, Alfonso Carreras Y, Al-Haddad C, Al-Hussaini HHY, Ali AM, Alia DB, Al-Jadiry MF, Al-Jumaily U, Alkatan HM, All-Eriksson C, Al-Mafrachi AARM, Almeida AA, Alsawidi KM, Al-Shaheen AASM, Al-Shammary EH, Amiruddin PO, Antonino R, Astbury NJ, Atalay HT, Atchaneeyasakul LO, Atsiaya R, Attaseth T, Aung TH, Ayala S, Baizakova B, Balaguer J, Balayeva R, Balwierz W, Barranco H, Bascaran C, Beck Popovic M, Benavides R, Benmiloud S, Bennani Guebessi N, Berete RC, Berry JL, Bhaduri A, Bhat S, Biddulph SJ, Biewald EM, Bobrova N, Boehme M, Boldt HC, Bonanomi MTBC, Bornfeld N, Bouda GC, Bouguila H, Boumedane A, Brennan RC, Brichard BG, Buaboonnam J, Calderon-Sotelo P, Calle Jara DA, Camuglia JE, Cano MR, Capra M, Cassoux N, Castela G, Castillo L, Catala-Mora J, Chantada GL, Chaudhry S, Chaugule SS, Chauhan A, Chawla B, Chernodrinska VS, Chiwanga FS, Chuluunbat T, Cieslik K, Cockcroft RL, Comsa C, Correa ZM, Correa Llano MG, Corson TW, Cowan-Lyn KE, Csoka M, Cui X, Da Gama IV, Dangboon W, Das A, Das S, Davanzo JM, Davidson A, De Potter P, Delgado KQ, Demirci H, Desjardins L, Diaz Coronado RY, Dimaras H, Dodgshun AJ, Donaldson C, Donato Macedo CR, Dragomir MD, Du Y, Du Bruyn M, Edison KS, Eka Sutyawan IW, El Kettani A, Elbahi AM, Elder JE, Elgalaly D, Elhaddad AM, Elhassan MMA, Elzembely MM, Essuman VA, Evina TGA, Fadoo Z, Fandino AC, Faranoush M, Fasina O, Fernandez DDPG, Fernandez-Teijeiro A, Foster A, Frenkel S, Fu LD, Fuentes-Alabi SL, Gallie BL, Gandiwa M, Garcia JL, Garcia Aldana D, Gassant PY, Geel JA, Ghassemi F, Giron AV, Gizachew Z, Goenz MA, Gold AS, Goldberg-Lavid M, Gole GA, Gomel N, Gonzalez E, Gonzalez Perez G, Gonzalez-Rodriguez L, Garcia Pacheco HN, Graells J, Green L, Gregersen PA, Grigorovski NDAK, Guedenon KM, Gunasekera DS, Gunduz AK, Gupta H, Gupta S, Hadjistilianou T, Hamel P, Hamid SA, Hamzah N, Hansen ED, Harbour JW, Hartnett ME, Hasanreisoglu M, Hassan S, Hassan S, Hederova S, Hernandez J, Hernandez LMC, Hessissen L, Hordofa DF, Huang LC, Hubbard GB, Hummlen M, Husakova K, Hussein Al-Janabi AN, Ida R, Ilic VR, Jairaj V, Jeeva I, Jenkinson H, Ji X, Jo DH, Johnson KP, Johnson WJ, Jones MM, Kabesha TBA, Kabore RL, Kaliki S, Kalinaki A, Kantar M, Kao LY, Kardava T, Kebudi R, Kepak T, Keren-Froim N, Khan ZJ, Khaqan HA, Khauv P, Kheir WJ, Khetan V, Khodabande A, Khotenashvili Z, Kim JW, Kim JH, Kiratli H, Kivela TT, Klett A, Komba Palet JEK, Krivaitiene D, Kruger M, Kulvichit K, Kuntorini MW, Kyara A, Lachmann ES, Lam CPS, Lam GC, Larson SA, Latinovic S, Laurenti KD, Le BHA, Lecuona K, Leverant AA, Li C, Limbu B, Long QB, Lopez JP, Lukamba RM, Lumbroso L, Luna-Fineman S, Lutfi D, Lysytsia L, Magrath GN, Mahajan A, Majeed AR, Maka E, Makan M, Makimbetov EK, Manda C, Martin Begue N, Mason L, Mason JO 3rd, Matende IO, Materin M, Mattosinho CCDS, Matua M, Mayet I, Mbumba FB, McKenzie JD, Medina-Sanson A, Mehrvar A, Mengesha AA, Menon V, Mercado GJVD, Mets MB, Midena E, Mishra DKC, Mndeme FG, Mohamedani AA, Mohammad MT, Moll AC, Montero MM, Morales RA, Moreira C, Mruthyunjaya P, Msina MS, Msukwa G, Mudaliar SS, Muma KI, Munier FL, Murgoi G, Murray TG, Musa KO, Mushtaq A, Mustak H, Muyen OM, Naidu G, Nair AG, Naumenko L, Ndoye Roth PA, Nency YM, Neroev V, Ngo H, Nieves RM, Nikitovic M, Nkanga ED, Nkumbe H, Nuruddin M, Nyaywa M, Obono-Obiang G, Oguego NC, Olechowski A, Oliver SCN, Osei-Bonsu P, Ossandon D, Paez-Escamilla MA, Pagarra H, Painter SL, Paintsil V, Paiva L, Pal BP, Palanivelu MS, Papyan R, Parrozzani R, Parulekar M, Pascual Morales CR, Paton KE, Pawinska-Wasikowska K, Pe'er J, Pena A, Peric S, Pham CTM, Philbert R, Plager DA, Pochop P, Polania RA, Polyakov VG, Pompe MT, Pons JJ, Prat D, Prom V, Purwanto I, Qadir AO, Qayyum S, Qian J, Rahman A, Rahman S, Rahmat J, Rajkarnikar P, Ramanjulu R, Ramasubramanian A, Ramirez-Ortiz MA, Raobela L, Rashid R, Reddy MA, Reich E, Renner LA, Reynders D, Ribadu D, Riheia MM, Ritter-Sovinz P, Rojanaporn D, Romero L, Roy SR, Saab RH, Saakyan S, Sabhan AH, Sagoo MS, Said AMA, Saiju R, Salas B, San Roman Pacheco S, Sanchez GL, Sayalith P, Scanlan TA, Schefler AC, Schoeman J, Sedaghat A, Seregard S, Seth R, Shah AS, Shakoor SA, Sharma MK, Sherief ST, Shetye NG, Shields CL, Siddiqui SN, Sidi Cheikh S, Silva S, Singh AD, Singh N, Singh U, Singha P, Sitorus RS, Skalet AH, Soebagjo HD, Sorochynska T, Ssali G, Stacey AW, Staffieri SE, Stahl ED, Stathopoulos C, Stirn Kranjc B, Stones DK, Strahlendorf C, Suarez MEC, Sultana S, Sun X, Sundy M, Superstein R, Supriyadi E, Surukrattanaskul S, Suzuki S, Svojgr K, Sylla F, Tamamyan G, Tan D, Tandili A, Tarrillo Leiva FF, Tashvighi M, Tateshi B, Tehuteru ES, Teixeira LF, Teh KH, Theophile T, Toledano H, Trang DL, Traore F, Trichaiyaporn S, Tuncer S, Tyau-Tyau H, Umar AB, Unal E, Uner OE, Urbak SF, Ushakova TL, Usmanov RH, Valeina S, van Hoefen Wijsard M, Varadisai A, Vasquez L, Vaughan LO, Veleva-Krasteva NV, Verma N, Victor AA, Viksnins M, Villacis Chafla EG, Vishnevskia-Dai V, Vora T, Wachtel AE, Wackernagel W, Waddell K, Wade PD, Wali AH, Wang YZ, Weiss A, Wilson MW, Wime ADC, Wiwatwongwana A, Wiwatwongwana D, Wolley Dod C, Wongwai P, Xiang D, Xiao Y, Yam JC, Yang H, Yanga JM, Yaqub MA, Yarovaya VA, Yarovoy AA, Ye H, Yousef YA, Yuliawati P, Zapata Lopez AM, Zein E, Zhang C, Zhang Y, Zhao J, Zheng X, Zhilyaeva K, Zia N, Ziko OAO, Zondervan M, Bowman R. Global Retinoblastoma Presentation and Analysis by National Income Level. JAMA Oncol. 2020 May 1;6(5):685-695. doi: 10.1001/jamaoncol.2019.6716. PMID 32105305
- [Result] Global Retinoblastoma Study Group. The Global Retinoblastoma Outcome Study: a prospective, cluster-based analysis of 4064 patients from 149 countries. Lancet Glob Health. 2022 Aug;10(8):e1128-e1140. doi: 10.1016/S2214-109X(22)00250-9. PMID 35839812